CLINICAL TRIAL: NCT05252871
Title: Assessment of Three Basic Progressive Lens Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Collaborators: Hoya Vision Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P21/IRB/065
Record Dates: First submitted 2022-01-03; First posted 2022-02-23 (Actual); Results first posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-07

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Progressive addition lens designs are unknown to participants, investigators, and outcomes assessors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Experimental: The specified PAL design wearers (Experimental): Subjects who have been already wearing any from specified design type of PAL
  Interventions: Device: Progressive Additional Lenses (PAL), pre calibrated and made of polymeric material with anti-reflection coating
- The other PAL design wearers (Active Comparator): Subjects who have been already wearing any from the other design type of PAL
  Interventions: Device: Progressive Additional Lenses (PAL), pre calibrated and made of polymeric material with anti-reflection coating

INTERVENTIONS:
Device: Progressive Additional Lenses (PAL), pre calibrated and made of polymeric material with anti-reflection coating — Subjects will be wearing three different PAL designs with different geometries of the optical progression.

SUMMARY:
This clinical trial investigates the differences between three different progressive addition lens designs. It is a non-invasive double-masked randomized clinical investigation. For this study, 80 participants will be recruited.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the preference, adaptability, and visual performance of three progressive lens designs. The difference in these lens designs is a variation of zone sizes for intermediate and near vision. The clinical trial helps manufacturers and eye care practitioners to give detailed suggestions to patients. Study participants will be experienced progressive addition lens wearers, which will be recruited by advertisements, by email, and with direct person-to-person solicitation. The study will be conducted at the Eye Care Institute at the Patient Care Center Western University of Health Sciences, Pomona, CA, 91766. For each participant, the study is completed in around two months and requires three separate visits.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45 to 70 years old.
* Visual Acuity: far & near monocular: cc ≥ 20/20 (decimal cc ≥ 1.0)
* Normal binocular vision (at distance & near: no strabismus on cover testing, aligning prism of less than 2Δ horizontally or vertically, stereoacuity of 2' or better at distance and near).
* Prescription is in the range:

  * Spherical power: less than +/-6.00 D
  * Cylindrical power: less than -2.75 D
  * Addition: 1.50 D - 2.50 D
  * Difference in power (spherical equivalent) between eyes: less than 2.00 D

Exclusion Criteria:

* Have never worn any progressive lens design.
* First prescription for progressive lenses.
* Prescription found during visit#1 varies from current prescription more than 0.50 D in any meridian.
* Currently wearing single vision lenses with accommodative support.
* Double vision or prismatic prescription in current glasses.
* Known ocular disease including strabismus, any pathology, any eye surgeries that may affect visual acuity.
* Use of systemic or ocular medications that are likely to affect vision.
* Balance problem/vertigo problem.
* Concurrent participation in other vision-related research.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Spors, Ph.D., Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Experimental: The Specified PAL Design Wearers | The Other PAL Design Wearers
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: The Specified PAL Design Wearers | The Other PAL Design Wearers | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 37 | 72
  >=65 years | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (7.11) | 55.6 (6.42) | 55.5 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 21 | 46
  Male | 15 | 19 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Adaptation to Progressive Lens Designs.
Description: Evaluate the adaptation to progressive lens designs through a "Satisfaction questionnaire" after 1 week of use of each of the 3 progressive addition lenses.
  Scale titles: Visual Quality Scale: A 5-point scale from a minimum value of 1 to a maximum score of 5. Higher scores mean better outcomes.
Time Frame: Entire study duration (approx. 4 weeks)
Population: For each participant, three pairs of progressive addition lenses were analyzed. Each pair was worn for one week.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Progressive Addition Lenses
Groups:
- Experimental: The Specified PAL Design Wearers, Wearing Pair 1: Subjects who have already been wearing the specified design type of PAL and wearing Pair 1 of the study lenses.
  Progressive Additional Lenses (PAL), pre-calibrated and made of polymeric material with anti-reflection coating: Subjects will be wearing three different PAL designs with different geometries of the optical progression.
- The Other PAL Design Wearers, Wearing Pair 1: Subjects who have been wearing any other design type of PAL and wearing Pair 1 of the study lenses.
  Progressive Additional Lenses (PAL), pre-calibrated and made of polymeric material with anti-reflection coating: Subjects will be wearing three different PAL designs with different geometries of the optical progression.
- Experimental: The Specified PAL Design Wearers, Wearing Pair 2: Subjects who have already been wearing the specified design type of PAL and wearing Pair 2 of the study lenses.
  Progressive Additional Lenses (PAL), pre-calibrated and made of polymeric material with anti-reflection coating: Subjects will be wearing three different PAL designs with different geometries of the optical progression.
- The Other PAL Design Wearers, Wearing Pair 2: Subjects who have been wearing any other design type of PAL and wearing Pair 2 of the study lenses.
  Progressive Additional Lenses (PAL), pre-calibrated and made of polymeric material with anti-reflection coating: Subjects will be wearing three different PAL designs with different geometries of the optical progression.
- Experimental: The Specified PAL Design Wearers, Wearing Pair 3: Subjects who have already been wearing the specified design type of PAL and wearing Pair 3 of the study lenses.
  Progressive Additional Lenses (PAL), pre-calibrated and made of polymeric material with anti-reflection coating: Subjects will be wearing three different PAL designs with different geometries of the optical progression.
- The Other PAL Design Wearers, Wearing Pair 3: Subjects who have been wearing any other design type of PAL and wearing Pair 3 of the study lenses.
  Progressive Additional Lenses (PAL), pre-calibrated and made of polymeric material with anti-reflection coating: Subjects will be wearing three different PAL designs with different geometries of the optical progression.
Arm/Group | Experimental: The Specified PAL Design Wearers, Wearing Pair 1 | The Other PAL Design Wearers, Wearing Pair 1 | Experimental: The Specified PAL Design Wearers, Wearing Pair 2 | The Other PAL Design Wearers, Wearing Pair 2 | Experimental: The Specified PAL Design Wearers, Wearing Pair 3 | The Other PAL Design Wearers, Wearing Pair 3
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Number analyzed (Progressive Addition Lenses) | 80 | 80 | 80 | 80 | 80 | 80
score on a scale | 4.125 (0.822) | 4.025 (1.05) | 3.875 (0.992) | 3.725 (0.987) | 4.300 (0.939) | 4.150 (0.864)

2. Secondary Outcome: Evaluate the Immediate Preference Among Progressive Lens Designs.
Description: Evaluate the immediate preference for progressive lens designs through a "Satisfaction questionnaire" directly after receiving the 3 progressive addition lenses.
  Scale titles: Visual Quality Scale: A 5-point scale from a minimum value of 1 to a maximum score of 5. Higher scores mean better outcomes.
Time Frame: Directly after receiving the lenses (approx. 15 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Progressive Addition Lenses
Arm/Group | Experimental: The Specified PAL Design Wearers, Wearing Pair 1 | The Other PAL Design Wearers, Wearing Pair 1 | Experimental: The Specified PAL Design Wearers, Wearing Pair 2 | The Other PAL Design Wearers, Wearing Pair 2 | Experimental: The Specified PAL Design Wearers, Wearing Pair 3 | The Other PAL Design Wearers, Wearing Pair 3
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Number analyzed (Progressive Addition Lenses) | 80 | 80 | 80 | 80 | 80 | 80
score on a scale | 4.550 (0.714) | 4.400 (0.709) | 4.625 (0.667) | 4.450 (0.783) | 4.625 (0.568) | 4.400 (0.672)

3. Secondary Outcome: Evaluate the Preference of Progressive Lens Designs.
Description: Evaluate the final preference of progressive lens designs after wearing each of the 3 PALs for one week.
  Scale title: Preference of Progressive Addition Lenses Scale: "Pair 1", "Pair 2, "Pair 3"
Time Frame: Entire study duration (approx. 4 weeks)
Population: For each participant, three pairs of progressive addition lenses were analyzed. Each pair was worn for one week.
Measure: Number; unit: participants
Units Other Than Participants: Progressive Addition Lenses
Arm/Group | Experimental: The Specified PAL Design Wearers, Wearing Pair 1 | The Other PAL Design Wearers, Wearing Pair 1 | Experimental: The Specified PAL Design Wearers, Wearing Pair 2 | The Other PAL Design Wearers, Wearing Pair 2 | Experimental: The Specified PAL Design Wearers, Wearing Pair 3 | The Other PAL Design Wearers, Wearing Pair 3
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
Number analyzed (Progressive Addition Lenses) | 80 | 80 | 80 | 80 | 80 | 80
participants | 11 | 16 | 10 | 9 | 19 | 15

ADVERSE EVENTS:
Time Frame: Through study completion, 6 months
Description: Each participant wore three pairs of progressive addition lenses for a total of three weeks. Potential adverse events included: Product Issues and Eye Disorders (reduced vision). The principal investigator was available for the study participants at any time during the study by phone and email to report adverse events. During the scheduled follow-up visits, participants were specifically asked for potential adverse events.
Arm/Group | Experimental: The Specified PAL Design Wearers, Wearing Pair 1 | The Other PAL Design Wearers, Wearing Pair 1 | Experimental: The Specified PAL Design Wearers, Wearing Pair 2 | The Other PAL Design Wearers, Wearing Pair 2 | Experimental: The Specified PAL Design Wearers, Wearing Pair 3 | The Other PAL Design Wearers, Wearing Pair 3
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40 | 0/40 | 0/40 | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
There are no limitations to be reported. The study went as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05252871/Prot_002.pdf
  • Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/71/NCT05252871/SAP_003.pdf